CLINICAL TRIAL: NCT04131426
Title: Evaluating the Effects of Dietary Supplementation With Remune on Cancer Associated Weight and Muscle Loss With and Without Exercise: A Randomized Pilot Feasibility Study.
Brief Title: Evaluating the Combined Intervention of Nutritional Supplementation (Remune) and Exercise in Patients With Cancer Cachexia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Smartfish AS (Industry)
Responsible Party: Principal Investigator, Richard Dunne, Assistant Professor - Department of Medicine , Hematology/Oncology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMLT19130
Record Dates: First submitted 2019-10-11; First posted 2019-10-18 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Cachexia; Cancer; Weight Loss; Lung Cancer; Gastrointestinal Cancer
Keywords: Cachexia; Cancer; Weight Loss; Exercise; Nutritional Supplement; Lung Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Cachexia; Neoplasms; Weight Loss; Lung Neoplasms; Gastrointestinal Neoplasms; Motor Activity | interventions — remune; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Remune dosed twice daily (Experimental): A nutritional supplement taken twice per day each day and standard care for your cancer as prescribed by your oncologist
  Interventions: Drug: Remune
- Remune dosed twice daily and daily exercise with EXCAP (Experimental): A nutritional supplement taken twice by day each day and a home-based exercise intervention as well as standard care for your cancer as prescribed by your oncologist
  Interventions: Drug: Remune; Other: EXCAP©®
- Usual Care (No Intervention): Usual standard care as prescribed by your oncologist

INTERVENTIONS:
Drug: Remune — Remune is intended for the dietary management of disease related malnutrition especially in patients with precachexia or cachexia due to cancer or COPD
  Arms: Remune dosed twice daily; Remune dosed twice daily and daily exercise with EXCAP
Other: EXCAP©® — EXCAP©® is a home-based low-to-moderate intensity program that employs a tailored walking prescription and total body resistance exercises
  Other Names: Exercise for Cancer Patients
  Arms: Remune dosed twice daily and daily exercise with EXCAP

SUMMARY:
The main purpose of this research study is to determine if the use of a nutritional supplement and exercise improve or worsen cachexia.

DETAILED DESCRIPTION:
In this study the investigator would like to better understand how cachexia may improve or worsen, and how exercise and nutritional supplements may impact this process. The investigator would like to see whether a nutritional supplement (Remune) with or without a walking and progressive resistance exercise program (EXCAP©®, Exercise for Cancer Patients) can improve symptoms in patients with lung or gastrointestinal cancers with weight loss and cachexia. The investigator would also like to find out if this nutritional supplement and exercise intervention improves physical performance, day-to-day function, quality of life, and how the supplement and/or exercise may affect different markers in the blood over time.

ELIGIBILITY:
Inclusion Criteria:

* Be over the age of 18 years and have a primary diagnosis of colorectal, esophageal, gastric, pancreatic, biliary tract cancer (includes cholangiocarcinoma, gallbladder cancer, and ampullary cancer), or Non-small cell lung cancer (NSCLC) with plans to initiate systemic chemotherapy, targeted therapy or immunotherapy within the next 4 weeks after enrollment.
* Have been diagnosed as having an unresectable cancer with no plans for surgical intervention during the active study period (12 weeks).
* Have an ECOG performance score of 0 or 1.
* Have a life expectancy of >3 months as determined by their primary oncologist.
* Have experienced at least 2% weight loss of the patient's reported previous body weight over the 6 months prior to enrollment.
* Have permission from primary oncologist to engage in low to moderate intensity exercise regimen.
* Be able to read English (since the assessment materials are in printed format).
* Be able to give written informed consent.

Exclusion Criteria:

* Have any of the following limitations: unable to perform low-to-moderate intensity exercise regimen.
* Have had major surgery (excluding diagnostic procedures like laparoscopy, EGD/EUS, esophageal stent placement) in the past 4 weeks.
* Be experiencing dysphagia that requires enteral or parenteral feeding for nutrition.
* Be enrolled on hospice at time of consent.
* Be engaged in an active exercise routine by being identified as in the Active or Maintenance Stage of exercise behavior as assessed by the 1-item Exercise Stages of Change Short Form (67).
* Use of nutritional supplements containing EPA/DHA within 2 weeks prior to screening
* Current Use of Vitamin D supplementation or St. John's wort that can influence efficacy and safety parameters. Chronic treatment (>12 weeks prior to screening) with multivitamin tablets is allowed (vitamin tablets must not contain more vitamin D than 150% of the recommended dietary allowance [RDA]).
* Known hypersensitivity or allergy to any of the study products. Specifically, patients allergic to milk, fish or shellfish will be excluded.
* Have AST/ALT >3x upper limit of normal (ULN) or >5xULN in those with liver metastases, Serum creatinine >2x ULN, Absolute Neutrophil Count <1,500/uL, Hemoglobin <9, Platelet count <75,000/uL at the time of baseline blood draw or any other Blood chemistry or hematology lab abnormalities that would exclude them from being able to receive standard chemotherapy or interventional clinical trial.
* Have uncontrolled Diabetes Mellitus as determined by primary oncologist or PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 months
  measured by adverse event severity and quantity
Adherance | 3 months
  Did 70% of subjects in the supplement arm consume 60% of supplement evening. Patients are asked to report the number of cartons of Remune consumed each day and how much they consumed
Recruitment and Retention | 3 months
  Recruitment of 45 patients (15 per arm) and at least 10 evaluable patients in each arm for retention rate of 66%

SECONDARY OUTCOMES:
Proportion of subjects that improve physical function- Walking | 3 months
  6 minute walk test distance; Participants are given a short warm up and cool down walking protocol in the test walking area in the University. During the 6-minute walk, participants will be asked to wear a sensor that will measure movement ability. The sensor is secured by an ergonomic belt around the participant's waist and allows for free body movement and comfort. Participants walk for a total of 6 minutes and cover as much distance as they can during this time. Upon completion of the test, the total distance walked is used to measure physical performance.
Proportion of subjects that improve physical function- Power | 3 months
  Power will be assessed by the Stair Climb Performance Test (SCPT) which is performed by having subjects safely ascend a flight of stairs (approximately 10 stairs total) as quick and as safely as possible with supervision. The subject can use the handrail as a safety precaution if deemed necessary by the patient, physician, coordinator, or exercise physiologist. Power is calculated by force (calculated by body mass and acceleration due to gravity) multiplied by the velocity (distance/time).
Proportion of subjects that improve physical function- Muscle Strength | 3 months
  Muscular strength will be assessed objectively using The Handgrip Dynamometer Test. The Handgrip Dynamometer Test is a grip strength test used to assess the maximal voluntary contraction generated by the arm muscles. The test is administered with the patient standing with the elbow joint angle held constant at 180 degrees and the medial distal humeral epicondyle held 2 inches from the torso. Trials will be performed in an alternating bilateral sequence, for a total of six attempts (three with each arm). The best score of the three hand-grip trials will be used for right and left limbs to calculate static strength.
Porportion of subjects with improved cachexia-related symptoms 3 months | 3 months
  The Functional Assessment of Anoreix/Cachexia Therapy subscale is a 39-item questionnaire that measures general aspects of quality of life as well as specific anorexia/cachexia-related concerns. This will be collected at pre- and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dunne, Principal Investigator — University of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States